CLINICAL TRIAL: NCT03174691
Title: The Early Luteal Progesterone Profile in IVF Patients Triggered With hCG
Brief Title: Early Luteal Progesterone Profile in IVF Patients Triggered With hCG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam National University (Other)
Collaborators: Mỹ Đức Hospital (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Doctor, Vietnam National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCKH/CGRH-09-2017
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: IVF patients triggered with hCG
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hormonal levels (Experimental): Collect blood samples Blood samples are collected on the following days after human chorionic gonadotropin (hCG) injection: Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 6
  Interventions: Diagnostic Test: Blood collection

INTERVENTIONS:
Diagnostic Test: Blood collection — A total of ten (10) blood samples (2ml/each) will be collected during the study.
  Blood samples will be collected on the following days for subsequent analysis of LH, Estradiol, hCG, progesterone and 17-Hydroxyprogesterone.

SUMMARY:
Until now very little information exists regarding the early luteal serum progesterone profile after Human chorionic gonadotropin (hCG) trigger. This pilot study will help characterize the serum progesterone, 17-hydroxyprogesterone profiles in IVF patients and correlate progesterone, 17-Hydroxyprogesterone levels to ovarian follicles obtained after stimulation with exogenous gonadotropins.

DETAILED DESCRIPTION:
The early luteal phase after IVF treatment is only scarcely studied. During IVF treatment the early luteinizing hormone (LH) activity deficit induced after ovarian stimulation with exogenous gonadotropins will be partly covered by the bolus of hCG used for triggering of final oocyte maturation due to the long half-life of hCG. In addition, the luteal phase will be covered by exogenous progesterone supplementation. After successful implantation the embryo itself will provide the supportive LH activity, securing the function of the corpora lutea. However, during the early luteal phase and peri-implantation, recent data suggest that an early-mid-luteal hCG/LH deficiency exists after hCG trigger during which the corpus luteum lacks an optimal stimulation. Furthermore, the early luteal progesterone profile in IVF differs significantly from the progesterone profile of the natural cycle, in which the peak is reached around the time of implantation. With this non-invasive trial, we wish to further explore the early luteal phase profiles of progesterone, 17-Hydroxyprogesterone and hCG in order to optimize current luteal phase support policies in IVF and hopefully increase ongoing pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Freeze all cycle after hCG trigger
* Age 18 - 38
* BMI < 28kg/m2
* Normal ovarian reserve, defined by Anti-Mullerian Hormone (AMH) > 1.25 ng/ml or Antral Follicle Count (AFC) ≥ 6 measured within two months prior to stimulation start
* Receiving gonadotrophin releasing hormone (GnRH) antagonist co-treatment during ovarian stimulation
* Agreement to participate in the study, and to disclose any medical events to the investigator. The subject must be willing and able to comply with the protocol requirements for the duration of the study.
* Have given written informed consent with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

* Previous poor response (≤ 3 oocytes) after high dose follicle stimulating hormone (FSH) stimulation
* Hyper-response defined as >20 follicles ≥ 14 mm
* Chronical medical conditions like Diabetes, Crohns disease, Thyroid disease, Hepatitis B and Sexually Transmitted Diseases Simultaneous participation in an interventional clinical trial.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of progesterone,17-Hydroxyprogesterone, LH, E2, and hCG during early luteal phase | In 6 days after human chorionic gonadotropin injection
  Blood samples are collected at ten points of time.

SECONDARY OUTCOMES:
Number of follicles ≥ 11 mm luteal phase | On the day of hCG injection
  Number of follicles are counted by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Principal Investigator — Research Center for Genetics and Reproductive Health Ho Chi Minh, Ho Chi Minh Vietnam
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vuong LN, Ho TM, Pham TD, Ho VNA, Andersen CY, Humaidan P. The early luteal hormonal profile in IVF patients triggered with hCG. Hum Reprod. 2020 Jan 1;35(1):157-166. doi: 10.1093/humrep/dez235. PMID 31967304